CLINICAL TRIAL: NCT05046132
Title: A Randomized, Double-Blind, 3-arm, Parallel Group, Placebo- and Positive-controlled Study to Investigate the Effects of Setmelanotide on QTc Interval in Healthy Subjects
Brief Title: Study of Setmelanotide Effects on QTc (Corrected QT) Interval in Healthy Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM-493-032; 263791 (Other: Paraxel)
Record Dates: First submitted 2021-07-30; First posted 2021-09-16 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — setmelanotide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Setmelanotide 2-7 mg + Placebo for Moxifloxacin (Experimental): Participants received titrated doses of 2-7 milligrams (mg) setmelanotide once daily by subcutaneous (SC) injection, starting with a dose of 2 mg from Days 1 to 7, 3 mg from Days 8 to 10, 5 mg from Days 11 to 13 and 7 mg from Days 14 to 16. Participants also received single oral dose of placebo matching moxifloxacin on Days 10 and 16.
  Interventions: Drug: Setmelanotide; Drug: Oral Placebo
- Group 2: Placebo for Setmelanotide + Moxifloxacin 400 mg + Placebo for Moxifloxacin (Active Comparator): Participants received placebo matching setmelanotide once daily by SC injection from Days 1 to 16. Participants also received a single oral dose of 400 mg moxifloxacin on Day 10 and a single oral dose of placebo matching moxifloxacin on Day 16.
  Interventions: Drug: Moxifloxacin; Drug: Oral Placebo; Drug: SC Placebo
- Group 3: Placebo for Setmelanotide + Placebo for Moxifloxacin + Moxifloxacin 400 mg (Active Comparator): Participants received placebo matching setmelanotide once daily by SC injection from Days 1 to 16. Participants also received a single oral dose of placebo matching moxifloxacin on Day 10 and a single oral dose of 400 mg moxifloxacin on Day 16.
  Interventions: Drug: Moxifloxacin; Drug: Oral Placebo; Drug: SC Placebo

INTERVENTIONS:
Drug: Setmelanotide — Administered once daily via SC injection.
  Arms: Group 1: Setmelanotide 2-7 mg + Placebo for Moxifloxacin
Drug: Moxifloxacin — Moxifloxacin capsules via oral administration.
  Arms: Group 2: Placebo for Setmelanotide + Moxifloxacin 400 mg + Placebo for Moxifloxacin; Group 3: Placebo for Setmelanotide + Placebo for Moxifloxacin + Moxifloxacin 400 mg
Drug: Oral Placebo — Placebo capsules via oral administration.
Drug: SC Placebo — Placebo via SC injection.
  Arms: Group 2: Placebo for Setmelanotide + Moxifloxacin 400 mg + Placebo for Moxifloxacin; Group 3: Placebo for Setmelanotide + Placebo for Moxifloxacin + Moxifloxacin 400 mg

SUMMARY:
This was a double-blind, randomized, placebo- and positive-controlled, parallel group, 3-arm study that assessed the potential for therapeutic and supratherapeutic concentrations of setmelanotide to affect the QTc corrected by the Fredericia method (QTcF) interval.

ELIGIBILITY:
Inclusion Criteria:

* Participant has body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2), inclusive.
* Participant is in good health, as confirmed by no clinically significant findings from medical history, physical examination, 12-lead Electrocardiogram (ECG), vital signs measurements, clinical laboratory evaluations, and liver function tests at Screening and Check-in.
* Female participants of childbearing potential must be confirmed non-pregnant and agree to use contraception.
* Male participants with female partners of childbearing potential must agree to use contraception. Male participants must also not donate sperm during and for 90 days following their participation in the study.
* Participant is a nonsmoker (for at least 3 months) with negative urinary cotinine test at Screening and agrees to abstain from alcohol, recreational drugs (including marijuana), and tobacco or nicotine-containing products for the duration of the study.
* Participant is able to comprehend and is willing to sign an informed consent form and abide by the study restrictions.

Exclusion Criteria:

* Participant has sustained systolic blood pressure (SBP) >150 millimeters of mercury (mmHg) or <90 mmHg or a diastolic blood pressure (DBP) >100 mmHg or <60 mmHg in the supine position at Screening or Day 1 of each study period, respectively.
* Participant has supine pulse rate of <45 beats per minute (bpm) or >100 bpm.
* Participant has abnormal screening ECG indicating a second- or third-degree atrioventricular block, or one or more of the following: QRS>110 millisecond (msec) , QTcF >450 msec for males and >470 msec for females, PR interval >200 msec.
* Participant has a history of risk factors for Torsades de Pointes (TdP), including unexplained syncope, diagnosis or family history of Brugada syndrome or long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, or hypomagnesaemia.
* Glomerular filtration rate (GFR) <60 milliliter per minute (mL/min) at Screening.
* Participant has significant dermatologic findings relating to melanoma or pre-melanoma skin lesions (excluding non-invasive basal or squamous cell lesion).
* Participant has history or close family history (parents or siblings) of melanoma or participant history of ocular-cutaneous albinism.
* Participant has significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator).
* Participant has suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening, a history of a suicide attempt in the last 20 years, or any suicidal behavior in the last month.
* Participant has participated in any clinical study with an investigational drug/device within 30 days (or 5 half-lives) prior to the first day of dosing.
* Participant was previously enrolled in a clinical study involving setmelanotide or any previous exposure to setmelanotide.
* Participant has inability to comply with once daily dosing (QD) injection regimen.
* Female participants who are breastfeeding or nursing.
* Participant has cognitive impairment that, in the investigator's opinion, precludes participation to the study.
* Participant is, in investigator's opinion, otherwise not suitable to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (1):
- Parexel Early Phase Clinical Unit (Los Angeles), Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 77 healthy participants aged 18 to 50 years, inclusive, were enrolled in the United States.
Pre-assignment Details: Participants were randomized 1:1:1 into Group 1, 2, or 3.
Period: Overall Study
Arm/Group | Group 1: Setmelanotide 2-7 mg + Placebo for Moxifloxacin | Group 2: Placebo for Setmelanotide + Moxifloxacin 400 mg + Placebo for Moxifloxacin | Group 3: Placebo for Setmelanotide + Placebo for Moxifloxacin + Moxifloxacin 400 mg
Started | 28 | 24 | 25
Received 2 mg Setmelanotide | 28 | 0 | 0
Received 3 mg Setmelanotide | 24 | 0 | 0
Received 5 mg Setmelanotide | 23 | 0 | 0
Received 7 mg Setmelanotide | 21 | 0 | 0
Completed | 21 | 23 | 25
Not Completed | 7 | 1 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Positive Covid19 Result. | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population included all participants who received at least one dose of study drug.
Groups:
- Group 1: Setmelanotide 2-7 mg + Placebo for Moxifloxacin: Participants received titrated doses of 2-7 mg setmelanotide once daily by SC injection, starting with a dose of 2 mg from Days 1 to 7, 3 mg from Days 8 to 10, 5 mg from Days 11 to 13 and 7 mg from Days 14 to 16. Participants also received single oral dose of placebo matching moxifloxacin on Days 10 and 16.
- Total: Total of all reporting groups
Arm/Group | Group 1: Setmelanotide 2-7 mg + Placebo for Moxifloxacin | Group 2: Placebo for Setmelanotide + Moxifloxacin 400 mg + Placebo for Moxifloxacin | Group 3: Placebo for Setmelanotide + Placebo for Moxifloxacin + Moxifloxacin 400 mg | Total
Number analyzed (Participants) | 28 | 24 | 25 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (6.47) | 36.1 (9.28) | 34.8 (8.60) | 34.2 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 12 | 33
  Male | 18 | 13 | 13 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 10 | 26
  Not Hispanic or Latino | 21 | 15 | 15 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 5 | 8 | 23
  White | 13 | 13 | 12 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Setmelanotide Concentration-related Placebo-corrected Change From Baseline (CHFB) in Fridericia's Correction (QTcF) at Day 10
Description: Continuous 12-lead digital electrocardiogram (ECG) recording was performed on Baseline and Day 10. ECG analysts were blinded to the treatment, timepoint and participant.
  QT interval was corrected for heart rate using QTcF. CHFB in QTcF was calculated at each timepoint.
Time Frame: Baseline and Day 10: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hours (hrs) postdose
Population: Pharmacokinetic (PK)/QTc Population included participants who were in both ECG & PK populations. PK Population included all participants who received at least 1 dose of setmelanotide or moxifloxacin & have at least 1 quantifiable concentration of setmelanotide or moxifloxacin. ECG Population included all participants in safety population with measurements at baseline as well as on-treatment with at least one post-dose timepoint with a valid value. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Groups:
- Group 1: Setmelanotide 3 mg: Participants received once daily setmelanotide 3 mg from Days 8 to 10, via SC injection.
- Group 3: Placebo: Participants received once daily placebo from Days 8 to 10, via SC injection.
Arm/Group | Group 1: Setmelanotide 3 mg | Group 3: Placebo
Number analyzed (Participants) | 23 | 25
milliseconds (msec)
  Predose | 1.9 (7.82) | -1.5 (5.25)
  0.5 hr Post dose | -3.6 (9.83) | -3.5 (8.16)
  1 hr Post dose | -2.9 (12.69) | -3.5 (5.87)
  1.5 hr Post dose | -3.0 (9.53) | -3.2 (7.44)
  2 hr Post dose | -1.0 (11.26) | -3.4 (5.70)
  2.5 hr Post dose: number analyzed (Participants) | 23 | 24
  2.5 hr Post dose | 1.2 (11.22) | -2.0 (8.92)
  3 hr Post dose: number analyzed (Participants) | 23 | 24
  3 hr Post dose | 2.1 (10.06) | -2.6 (6.75)
  4 hr Post dose | 2.0 (9.76) | -2.4 (8.09)
  5 hr Post dose: number analyzed (Participants) | 23 | 24
  5 hr Post dose | 2.4 (9.38) | 0.2 (8.99)
  6 hr Post dose: number analyzed (Participants) | 23 | 24
  6 hr Post dose | -0.4 (9.71) | -1.8 (6.88)
  7 hr Post dose: number analyzed (Participants) | 23 | 24
  7 hr Post dose | 1.0 (8.02) | -1.3 (7.36)
  8 hr Post dose: number analyzed (Participants) | 23 | 24
  8 hr Post dose | 2.6 (9.11) | -0.3 (7.93)
  9 hr Post dose: number analyzed (Participants) | 23 | 22
  9 hr Post dose | 4.1 (7.84) | -2.0 (6.58)
  10 hr Post dose: number analyzed (Participants) | 23 | 24
  10 hr Post dose | 5.0 (8.14) | -0.9 (9.96)
  12 hr Post dose: number analyzed (Participants) | 23 | 24
  12 hr Post dose | 1.9 (9.25) | 3.4 (8.65)
  16 hr Post dose: number analyzed (Participants) | 22 | 24
  16 hr Post dose | 1.7 (7.46) | -1.0 (7.64)
  24 hr Post dose: number analyzed (Participants) | 21 | 22
  24 hr Post dose | -0.7 (13.32) | 1.6 (8.28)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 3 mg vs Group 3: Placebo; The C-QTc analysis was performed with a non-linear model. The mean of placebo-corrected CHFB in QTcF at maximum concentration (Cmax) geometric mean of therapeutic dose (3 mg QD) was estimated with bias-corrected 90% CI by nonparametric bootstrap methods; Test type: Other; Mean of Placebo-corrected CHFB = 3.70, 90% CI 2-sided [1.23 to 6.17], Standard Error of Mean 1.48

2. Primary Outcome: Setmelanotide Concentration-related Placebo-corrected CHFB in QTcF at Day 16
Description: Continuous 12-lead digital ECG recording was performed on Baseline and Day 16. ECG analysts were blinded to the treatment, timepoint and participant.
  QT interval was corrected for heart rate using QTcF. CHFB in QTcF was calculated at each timepoint.
Time Frame: Baseline and Day 16: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: PK/QTc Population included participants who were in both ECG & PK populations. PK Population included all participants who received at least 1 dose of setmelanotide or moxifloxacin and have at least one quantifiable concentration of setmelanotide or moxifloxacin. ECG Population included all participants in safety population with measurements at baseline as well as on-treatment with at least one post-dose timepoint with a valid value. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Group 1: Setmelanotide 7 mg: Participants received once daily setmelanotide 7 mg from Days 14 to 16, via SC injection.
- Group 2: Placebo: Participants received once daily placebo from Days 14 to 16, via SC injection.
Arm/Group | Group 1: Setmelanotide 7 mg | Group 2: Placebo
Number analyzed (Participants) | 21 | 23
msec
  Predose | 4.5 (6.49) | -2.3 (8.24)
  0.5 hr Post dose | 1.0 (8.83) | -5.2 (6.97)
  1 hr Post dose | 1.6 (9.18) | -4.3 (8.20)
  1.5 hr Post dose: number analyzed (Participants) | 21 | 21
  1.5 hr Post dose | 0.3 (10.42) | -2.9 (8.64)
  2 hr Post dose: number analyzed (Participants) | 21 | 20
  2 hr Post dose | 2.2 (10.94) | -2.0 (8.96)
  2.5 hr Post dose: number analyzed (Participants) | 21 | 22
  2.5 hr Post dose | 2.7 (11.61) | -2.5 (9.09)
  3 hr Post dose: number analyzed (Participants) | 21 | 21
  3 hr Post dose | 4.3 (11.34) | -2.0 (8.07)
  4 hr Post dose: number analyzed (Participants) | 21 | 22
  4 hr Post dose | 3.6 (9.88) | -2.5 (6.37)
  5 hr Post dose: number analyzed (Participants) | 20 | 21
  5 hr Post dose | 4.7 (9.41) | -0.5 (6.42)
  6 hr Post dose: number analyzed (Participants) | 20 | 23
  6 hr Post dose | 2.8 (9.64) | -2.4 (7.28)
  7 hr Post dose | 1.5 (11.14) | -2.0 (6.31)
  8 hr Post dose | 2.8 (10.02) | -2.6 (8.27)
  9 hr Post dose: number analyzed (Participants) | 21 | 22
  9 hr Post dose | 6.1 (8.72) | -1.2 (7.00)
  10 hr Post dose: number analyzed (Participants) | 21 | 21
  10 hr Post dose | 6.5 (6.64) | -2.5 (7.14)
  12 hr Post dose: number analyzed (Participants) | 21 | 21
  12 hr Post dose | 5.8 (7.96) | -0.4 (5.99)
  16 hr Post dose: number analyzed (Participants) | 20 | 22
  16 hr Post dose | 1.4 (7.77) | -2.6 (9.30)
  24 hr Post dose: number analyzed (Participants) | 20 | 21
  24 hr Post dose | 1.0 (11.26) | -5.6 (9.67)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 7 mg vs Group 2: Placebo; The C-QTc analysis was performed with a non-linear model. The mean of placebo-corrected CHFB in QTcF at Cmax geometric mean of therapeutic dose (7 mg QD) was estimated with bias-corrected 90% CI by nonparametric bootstrap methods; Test type: Other; Mean of Placebo-corrected CHFB = 4.67, 90% CI 2-sided [1.70 to 7.64]

3. Secondary Outcome: Placebo-corrected CHFB in Heart Rate (HR) After Administration of SC Setmelanotide or Oral Moxifloxacin at Day 10
Description: The CHFB in HR was analyzed using an analysis of variance model (ANOVA) including treatment, time and their interaction as main factors and structuring the residual matrix in order to account for the repeated measurement pattern of the data. HR was considered as covariate. Placebo corrected values were reported in the inferential statistics.
Time Frame: Baseline and Day 10: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hours (hrs) postdose
Population: ECG population with available data was analyzed. ECG data was collected on Day 10 where participants received setmelanotide 3 mg.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Groups:
- Group 1: Setmelanotide 3 mg: Participants received once daily setmelanotide 3 mg QD from Days 8 to 10, via SC injection.
- Group 2: Moxifloxacin 400 mg: Participants received a single oral dose of 400 mg moxifloxacin on Day 10.
Arm/Group | Group 1: Setmelanotide 3 mg | Group 2: Moxifloxacin 400 mg
Number analyzed (Participants) | 23 | 23
beats per minute (bpm)
  Pre dose | 2.3 (9.65) | -0.3 (7.31)
  0.5 hr Post dose | -2.0 (9.58) | 0.9 (6.39)
  1 hr Post dose | -2.7 (11.67) | 1.3 (5.79)
  1.5 hr Post dose: number analyzed (Participants) | 23 | 21
  1.5 hr Post dose | -0.2 (13.13) | 2.0 (5.51)
  2 hr Post dose: number analyzed (Participants) | 23 | 21
  2 hr Post dose | -2.1 (10.94) | 0.0 (6.77)
  2.5 hr Post dose | -1.8 (9.31) | 1.7 (6.33)
  3 hr Post dose | 0.2 (10.70) | -0.4 (8.47)
  4 hr Post dose | -1.2 (7.91) | -0.6 (6.26)
  5 hr Post dose | 0.6 (7.51) | 3.1 (7.36)
  6 hr Post dose | -1.3 (7.66) | 3.6 (5.97)
  7 hr Post dose | -2.9 (6.45) | 0.9 (4.74)
  8 hr Post dose | -2.2 (5.93) | 2.4 (7.04)
  9 hr Post dose: number analyzed (Participants) | 23 | 22
  9 hr Post dose | -1.3 (6.34) | 1.3 (6.27)
  10 hr Post dose: number analyzed (Participants) | 23 | 22
  10 hr Post dose | -0.8 (5.82) | 0.9 (5.33)
  12 hr Post dose: number analyzed (Participants) | 23 | 22
  12 hr Post dose | -2.8 (7.49) | 3.3 (6.03)
  16 hr Post dose: number analyzed (Participants) | 22 | 22
  16 hr Post dose | 1.7 (6.93) | 1.9 (7.00)
  24 hr Post dose: number analyzed (Participants) | 21 | 22
  24 hr Post dose | 2.1 (6.04) | 1.3 (5.37)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 3 mg; Pre-dose; Test type: Other; LS Mean = 2.5, 90% CI 2-sided [-0.6 to 5.6]
Statistical Analysis 2: Comparison: Group 1: Setmelanotide 3 mg; 0.5 hr Post dose; Test type: Other; LS Mean = 0.1, 90% CI 2-sided [-3.0 to 3.1]
Statistical Analysis 3: Comparison: Group 1: Setmelanotide 3 mg; 1 hr Post dose; Test type: Other; LS Mean = 0.1, 90% CI 2-sided [-2.8 to 3.0]
Statistical Analysis 4: Comparison: Group 1: Setmelanotide 3 mg; 1.5 hr Post dose; Test type: Other; LS Mean = 1.6, 90% CI 2-sided [-1.8 to 5.1]
Statistical Analysis 5: Comparison: Group 1: Setmelanotide 3 mg; 2 hr Post dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-2.8 to 4.1]
Statistical Analysis 6: Comparison: Group 1: Setmelanotide 3 mg; 2.5 hr Post dose; Test type: Other; LS Mean = 0.2, 90% CI 2-sided [-2.9 to 3.4]
Statistical Analysis 7: Comparison: Group 1: Setmelanotide 3 mg; 3 hr Post dose; Test type: Other; LS Mean = 2.2, 90% CI 2-sided [-1.4 to 5.7]
Statistical Analysis 8: Comparison: Group 1: Setmelanotide 3 mg; 4 hr Post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-2.9 to 2.7]
Statistical Analysis 9: Comparison: Group 1: Setmelanotide 3 mg; 5 hr Post dose; Test type: Other; LS Mean = -0.2, 90% CI 2-sided [-3.1 to 2.7]
Statistical Analysis 10: Comparison: Group 1: Setmelanotide 3 mg; 6 hr Post dose; Test type: Other; LS Mean = -0.8, 90% CI 2-sided [-3.8 to 2.3]
Statistical Analysis 11: Comparison: Group 1: Setmelanotide 3 mg; 7 hr Post dose; Test type: Other; LS Mean = -2.8, 90% CI 2-sided [-5.5 to -0.1]
Statistical Analysis 12: Comparison: Group 1: Setmelanotide 3 mg; 8 hr Post dose; Test type: Other; LS Mean = -1.6, 90% CI 2-sided [-4.5 to 1.3]
Statistical Analysis 13: Comparison: Group 1: Setmelanotide 3 mg; 9 hr Post dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-2.5 to 3.0]
Statistical Analysis 14: Comparison: Group 1: Setmelanotide 3 mg; 10 hr Post dose; Test type: Other; LS Mean = 0.2, 90% CI 2-sided [-2.3 to 2.7]
Statistical Analysis 15: Comparison: Group 1: Setmelanotide 3 mg; 12 hr Post dose; Test type: Other; LS Mean = -3.0, 90% CI 2-sided [-5.9 to -0.1]
Statistical Analysis 16: Comparison: Group 1: Setmelanotide 3 mg; 16 hr Post dose; Test type: Other; LS Mean = -2.0, 90% CI 2-sided [-5.1 to 1.0]
Statistical Analysis 17: Comparison: Group 1: Setmelanotide 3 mg; 24 hr Post dose; Test type: Other; LS Mean = 1.1, 90% CI 2-sided [-1.6 to 3.8]
Statistical Analysis 18: Comparison: Group 2: Moxifloxacin 400 mg; Pre-dose; Test type: Other; LS Mean = 1.4, 90% CI 2-sided [-1.7 to 4.5]
Statistical Analysis 19: Comparison: Group 2: Moxifloxacin 400 mg; 0.5 hr Post dose; Test type: Other; LS Mean = 1.7, 90% CI 2-sided [-1.4 to 4.7]
Statistical Analysis 20: Comparison: Group 2: Moxifloxacin 400 mg; 1 hr Post dose; Test type: Other; LS Mean = 1.9, 90% CI 2-sided [-1.0 to 4.8]
Statistical Analysis 21: Comparison: Group 2: Moxifloxacin 400 mg; 1.5 hr Post dose; Test type: Other; LS Mean = 2.6, 90% CI 2-sided [-0.9 to 6.0]
Statistical Analysis 22: Comparison: Group 2: Moxifloxacin 400 mg; 2 hr Post dose; Test type: Other; LS Mean = 1.3, 90% CI 2-sided [-2.1 to 4.8]
Statistical Analysis 23: Comparison: Group 2: Moxifloxacin 400 mg; 2.5 hr Post dose; Test type: Other; LS Mean = 1.7, 90% CI 2-sided [-1.4 to 4.9]
Statistical Analysis 24: Comparison: Group 2: Moxifloxacin 400 mg; 3 hr Post dose; Test type: Other; LS Mean = 1.6, 90% CI 2-sided [-1.9 to 5.1]
Statistical Analysis 25: Comparison: Group 2: Moxifloxacin 400 mg; 4 hr Post dose; Test type: Other; LS Mean = 1.4, 90% CI 2-sided [-1.4 to 4.2]
Statistical Analysis 26: Comparison: Group 2: Moxifloxacin 400 mg; 5 hr Post dose; Test type: Other; LS Mean = 2.7, 90% CI 2-sided [-0.2 to 5.7]
Statistical Analysis 27: Comparison: Group 2: Moxifloxacin 400 mg; 6 hr Post dose; Test type: Other; LS Mean = 4.4, 90% CI 2-sided [1.4 to 7.5]
Statistical Analysis 28: Comparison: Group 2: Moxifloxacin 400 mg; 7 hr Post dose; Test type: Other; LS Mean = 2.8, 90% CI 2-sided [0.1 to 5.5]
Statistical Analysis 29: Comparison: Group 2: Moxifloxacin 400 mg; 8 hr Post dose; Test type: Other; LS Mean = 4.1, 90% CI 2-sided [1.2 to 7.0]
Statistical Analysis 30: Comparison: Group 2: Moxifloxacin 400 mg; 9 hr Post dose; Test type: Other; LS Mean = 3.6, 90% CI 2-sided [0.8 to 6.3]
Statistical Analysis 31: Comparison: Group 2: Moxifloxacin 400 mg; 10 hr Post dose; Test type: Other; LS Mean = 3.3, 90% CI 2-sided [0.8 to 5.8]
Statistical Analysis 32: Comparison: Group 2: Moxifloxacin 400 mg; 12 hr Post dose; Test type: Other; LS Mean = 2.6, 90% CI 2-sided [-0.3 to 5.5]
Statistical Analysis 33: Comparison: Group 2: Moxifloxacin 400 mg; 16 hr Post dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-2.7 to 3.4]
Statistical Analysis 34: Comparison: Group 2: Moxifloxacin 400 mg; 24 hr Post dose; Test type: Other; LS Mean = 1.7, 90% CI 2-sided [-1.0 to 4.4]

4. Secondary Outcome: Placebo-corrected CHFB in HR After Administration of SC Setmelanotide or Oral Moxifloxacin at Day 16
Description: The CHFB in HR was analysed using an ANOVA including treatment, time and their interaction as main factors and structuring the residual matrix in order to account for the repeated measurement pattern of the data. HR was considered as covariate.
Time Frame: Baseline and Day 16: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: ECG population with available data was analyzed. ECG data was collected on Day 16, where participants received setmelanotide 7 mg.
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- Group 3: Moxifloxacin 400 mg: Participants received a single oral dose of 400 mg moxifloxacin on Day 16.
Arm/Group | Group 1: Setmelanotide 7 mg | Group 3: Moxifloxacin 400 mg
Number analyzed (Participants) | 21 | 25
bpm
  Pre dose: number analyzed (Participants) | 21 | 24
  Pre dose | 3.4 (7.41) | -0.3 (4.95)
  0.5 hr Post dose | -1.7 (9.57) | -0.1 (6.35)
  1 hr Post dose | -2.2 (10.61) | 0.1 (5.96)
  1.5 hr Post dose: number analyzed (Participants) | 21 | 24
  1.5 hr Post dose | -1.5 (10.35) | 1.5 (5.78)
  2 hr Post dose | -3.0 (7.19) | 0.5 (5.14)
  2.5 hr Post dose | -0.8 (7.24) | 0.4 (6.49)
  3 hr Post dose | -0.2 (7.11) | 2.1 (5.44)
  4 hr Post dose: number analyzed (Participants) | 20 | 25
  4 hr Post dose | 1.5 (6.90) | 2.0 (5.18)
  5 hr Post dose: number analyzed (Participants) | 20 | 25
  5 hr Post dose | 3.5 (7.84) | 3.4 (5.76)
  6 hr Post dose: number analyzed (Participants) | 20 | 25
  6 hr Post dose | 3.9 (9.21) | 0.7 (5.66)
  7 hr Post dose | 1.2 (6.71) | 3.3 (7.68)
  8 hr Post dose: number analyzed (Participants) | 21 | 23
  8 hr Post dose | 0.8 (7.13) | 2.8 (4.71)
  9 hr Post dose: number analyzed (Participants) | 21 | 23
  9 hr Post dose | 1.5 (7.30) | 1.6 (6.59)
  10 hr Post dose | 2.1 (7.82) | 2.8 (5.16)
  12 hr Post dose: number analyzed (Participants) | 21 | 24
  12 hr Post dose | 0.6 (8.00) | 3.0 (3.86)
  16 hr Post dose: number analyzed (Participants) | 20 | 24
  16 hr Post dose | 3.0 (6.98) | 3.3 (4.75)
  24 hr Post dose: number analyzed (Participants) | 20 | 23
  24 hr Post dose | 6.2 (7.41) | 0.4 (6.39)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 7 mg; Pre dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-2.8 to 3.4]
Statistical Analysis 2: Comparison: Group 1: Setmelanotide 7 mg; 0.5 hr Post dose; Test type: Other; LS Mean = -2.1, 90% CI 2-sided [-5.3 to 1.0]
Statistical Analysis 3: Comparison: Group 1: Setmelanotide 7 mg; 1 hr Post dose; Test type: Other; LS Mean = -1.6, 90% CI 2-sided [-4.7 to 1.4]
Statistical Analysis 4: Comparison: Group 1: Setmelanotide 7 mg; 1.5 hr Post dose; Test type: Other; LS Mean = -2.2, 90% CI 2-sided [-5.3 to 1.0]
Statistical Analysis 5: Comparison: Group 1: Setmelanotide 7 mg; 2 hr Post dose; Test type: Other; LS Mean = -3.3, 90% CI 2-sided [-6.3 to -0.3]
Statistical Analysis 6: Comparison: Group 1: Setmelanotide 7 mg; 2.5 hr Post dose; Test type: Other; LS Mean = -1.2, 90% CI 2-sided [-4.1 to 1.7]
Statistical Analysis 7: Comparison: Group 1: Setmelanotide 7 mg; 3 hr Post dose; Test type: Other; LS Mean = -1.3, 90% CI 2-sided [-4.2 to 1.7]
Statistical Analysis 8: Comparison: Group 1: Setmelanotide 7 mg; 4 hr Post dose; Test type: Other; LS Mean = -0.6, 90% CI 2-sided [-3.6 to 2.5]
Statistical Analysis 9: Comparison: Group 1: Setmelanotide 7 mg; 5 hr Post dose; Test type: Other; LS Mean = -1.0, 95% CI 2-sided [-4.1 to 2.1]
Statistical Analysis 10: Comparison: Group 1: Setmelanotide 7 mg; 6 hr Post dose; Test type: Other; LS Mean = 0.4, 90% CI 2-sided [-2.7 to 3.5]
Statistical Analysis 11: Comparison: Group 1: Setmelanotide 7 mg; 7 hr Post dose; Test type: Other; LS Mean = -2.5, 90% CI 2-sided [-5.5 to 0.5]
Statistical Analysis 12: Comparison: Group 1: Setmelanotide 7 mg; 8 hr Post dose; Test type: Other; LS Mean = -2.2, 90% CI 2-sided [-5.2 to 0.8]
Statistical Analysis 13: Comparison: Group 1: Setmelanotide 7 mg; 9 hr Post dose; Test type: Other; LS Mean = -0.9, 90% CI 2-sided [-4.3 to 2.6]
Statistical Analysis 14: Comparison: Group 1: Setmelanotide 7 mg; 10 hr Post dose; Test type: Other; LS Mean = -0.2, 90% CI 2-sided [-3.6 to 3.2]
Statistical Analysis 15: Comparison: Group 1: Setmelanotide 7 mg; 12 hr Post dose; Test type: Other; LS Mean = -2.2, 90% CI 2-sided [-5.5 to 1.0]
Statistical Analysis 16: Comparison: Group 1: Setmelanotide 7 mg; 16 hr Post dose; Test type: Other; LS Mean = -1.9, 90% CI 2-sided [-5.4 to 1.7]
Statistical Analysis 17: Comparison: Group 1: Setmelanotide 7 mg; 24 hr Post dose; Test type: Other; LS Mean = 2.6, 90% CI 2-sided [-1.2 to 6.3]
Statistical Analysis 18: Comparison: Group 3: Moxifloxacin 400 mg; Pre-dose; Test type: Other; LS Mean = -2.1, 90% CI 2-sided [-5.1 to 0.8]
Statistical Analysis 19: Comparison: Group 3: Moxifloxacin 400 mg; 0.5 hr Post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-3.1 to 3.0]
Statistical Analysis 20: Comparison: Group 3: Moxifloxacin 400 mg; 1 hr Post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-3.0 to 2.9]
Statistical Analysis 21: Comparison: Group 3: Moxifloxacin 400 mg; 1.5 hr Post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-3.1 to 3.0]
Statistical Analysis 22: Comparison: Group 3: Moxifloxacin 400 mg; 2 hr Post dose; Test type: Other; LS Mean = -0.9, 90% CI 2-sided [-3.8 to 2.0]
Statistical Analysis 23: Comparison: Group 3: Moxifloxacin 400 mg; 2.5 hr Post dose; Test type: Other; LS Mean = 0.2, 90% CI 2-sided [-2.5 to 3.0]
Statistical Analysis 24: Comparison: Group 3: Moxifloxacin 400 mg; 3 hr Post dose; Test type: Other; LS Mean = 0.9, 90% CI 2-sided [-1.9 to 3.7]
Statistical Analysis 25: Comparison: Group 3: Moxifloxacin 400 mg; 4 hr Post dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-2.2 to 3.7]
Statistical Analysis 26: Comparison: Group 3: Moxifloxacin 400 mg; 5 hr Post dose; Test type: Other; LS Mean = 0.1, 90% CI 2-sided [-2.8 to 3.1]
Statistical Analysis 27: Comparison: Group 3: Moxifloxacin 400 mg; 6 hr Post dose; Test type: Other; LS Mean = -0.9, 90% CI 2-sided [-3.9 to 2.0]
Statistical Analysis 28: Comparison: Group 3: Moxifloxacin 400 mg; 7 hr Post dose; Test type: Other; LS Mean = -0.2, 90% CI 2-sided [-3.1 to 2.7]
Statistical Analysis 29: Comparison: Group 3: Moxifloxacin 400 mg; 8 hr Post dose; Test type: Other; LS Mean = 0.2, 90% CI 2-sided [-2.7 to 3.1]
Statistical Analysis 30: Comparison: Group 3: Moxifloxacin 400 mg; 9 hr Post dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-2.7 to 4.0]
Statistical Analysis 31: Comparison: Group 3: Moxifloxacin 400 mg; 10 hr Post dose; Test type: Other; LS Mean = 0.9, 90% CI 2-sided [-2.3 to 4.1]
Statistical Analysis 32: Comparison: Group 3: Moxifloxacin 400 mg; 12 hr Post dose; Test type: Other; LS Mean = -0.4, 90% CI 2-sided [-3.5 to 2.8]
Statistical Analysis 33: Comparison: Group 3: Moxifloxacin 400 mg; 16 hr Post dose; Test type: Other; LS Mean = -0.4, 90% CI 2-sided [-3.8 to 3.0]
Statistical Analysis 34: Comparison: Group 3: Moxifloxacin 400 mg; 24 hr Post dose; Test type: Other; LS Mean = -1.6, 90% CI 2-sided [-5.1 to 2.0]

5. Secondary Outcome: Placebo-corrected CHFB in QTcF Intervals After Administration of SC Setmelanotide or Oral Moxifloxacin at Day 10
Description: The CHFB in QTcF was analyzed using an ANOVA including treatment, time and their interaction as main factors and structuring the residual matrix in order to account for the repeated measurement pattern of the data. HR was considered as covariate.
Time Frame: Baseline and Day 10: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: ECG population with available data was analyzed. ECG data was collected on Day 10, where participants received setmelanotide 3 mg.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Group 1: Setmelanotide 3 mg | Group 2: Moxifloxacin 400 mg
Number analyzed (Participants) | 23 | 23
msec
  Pre dose | 1.9 (7.82) | 1.5 (7.76)
  0.5 hr Post dose | -3.6 (9.83) | -5.3 (8.75)
  1 hr Post dose | -2.9 (12.69) | -3.7 (9.39)
  1.5 hr Post dose: number analyzed (Participants) | 23 | 21
  1.5 hr Post dose | -3.0 (9.53) | 0.9 (8.56)
  2 hr Post dose: number analyzed (Participants) | 23 | 21
  2 hr Post dose | -1.0 (11.26) | 2.0 (8.74)
  2.5 hr Post dose | 1.2 (11.22) | 4.9 (8.75)
  3 hr Post dose | 2.1 (10.06) | 4.9 (7.39)
  4 hr Post dose | 2.0 (9.76) | 6.3 (8.63)
  5 hr Post dose: number analyzed (Participants) | 23 | 22
  5 hr Post dose | 2.4 (9.38) | 8.1 (8.42)
  6 hr Post dose | -0.4 (9.71) | 6.0 (6.61)
  7 hr Post dose | 1.0 (8.02) | 5.1 (8.39)
  8 hr Post dose | 2.6 (9.11) | 4.4 (8.18)
  9 hr Post dose: number analyzed (Participants) | 23 | 22
  9 hr Post dose | 4.1 (7.84) | 5.0 (10.47)
  10 hr Post dose: number analyzed (Participants) | 23 | 22
  10 hr Post dose | 5.0 (8.14) | 6.2 (6.85)
  12 hr Post dose: number analyzed (Participants) | 23 | 22
  12 hr Post dose | 1.9 (9.25) | 8.7 (4.84)
  16 hr Post dose: number analyzed (Participants) | 22 | 22
  16 hr Post dose | 1.7 (7.46) | 5.9 (8.09)
  24 hr Post dose: number analyzed (Participants) | 21 | 22
  24 hr Post dose | -0.7 (13.32) | 6.6 (8.00)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 3 mg; Pre dose; Test type: Other; LS Mean = 3.5, 90% CI 2-sided [0.1 to 6.8]
Statistical Analysis 2: Comparison: Group 1: Setmelanotide 3 mg; 0.5 hr Post dose; Test type: Other; LS Mean = 0.8, 90% CI 2-sided [-3.0 to 4.6]
Statistical Analysis 3: Comparison: Group 1: Setmelanotide 3 mg; 1 hr Post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-4.1 to 3.9]
Statistical Analysis 4: Comparison: Group 1: Setmelanotide 3 mg; 1.5 hr Post dose; Test type: Other; LS Mean = 0.9, 90% CI 2-sided [-2.7 to 4.4]
Statistical Analysis 5: Comparison: Group 1: Setmelanotide 3 mg; 2 hr Post dose; Test type: Other; LS Mean = 3.0, 90% CI 2-sided [-0.6 to 6.6]
Statistical Analysis 6: Comparison: Group 1: Setmelanotide 3 mg; 2.5 hr Post dose; Test type: Other; LS Mean = 3.5, 90% CI 2-sided [-0.3 to 7.4]
Statistical Analysis 7: Comparison: Group 1: Setmelanotide 3 mg; 3 hr Post dose; Test type: Other; LS Mean = 4.6, 90% CI 2-sided [1.2 to 8.1]
Statistical Analysis 8: Comparison: Group 1: Setmelanotide 3 mg; 4 hr Post dose; Test type: Other; LS Mean = 5.2, 90% CI 2-sided [1.5 to 8.9]
Statistical Analysis 9: Comparison: Group 1: Setmelanotide 3 mg; 5 hr Post dose; Test type: Other; LS Mean = 2.0, 90% CI 2-sided [-1.7 to 5.8]
Statistical Analysis 10: Comparison: Group 1: Setmelanotide 3 mg; 6 hr Post dose; Test type: Other; LS Mean = 1.7, 90% CI 2-sided [-1.6 to 5.1]
Statistical Analysis 11: Comparison: Group 1: Setmelanotide 3 mg; 7 hr Post dose; Test type: Other; LS Mean = 2.3, 90% CI 2-sided [-1.1 to 5.7]
Statistical Analysis 12: Comparison: Group 1: Setmelanotide 3 mg; 8 hr Post dose; Test type: Other; LS Mean = 2.4, 90% CI 2-sided [-1.4 to 6.2]
Statistical Analysis 13: Comparison: Group 1: Setmelanotide 3 mg; 9 hr Post dose; Test type: Other; LS Mean = 4.4, 90% CI 2-sided [0.9 to 7.8]
Statistical Analysis 14: Comparison: Group 1: Setmelanotide 3 mg; 10 hr Post dose; Test type: Other; LS Mean = 3.8, 90% CI 2-sided [0.3 to 7.4]
Statistical Analysis 15: Comparison: Group 1: Setmelanotide 3 mg; 12 hr Post dose; Test type: Other; LS Mean = -0.8, 90% CI 2-sided [-4.2 to 2.7]
Statistical Analysis 16: Comparison: Group 1: Setmelanotide 3 mg; 16 hr Post dose; Test type: Other; LS Mean = 3.6, 90% CI 2-sided [0.1 to 7.0]
Statistical Analysis 17: Comparison: Group 1: Setmelanotide 3 mg; 24 hr Post dose; Test type: Other; LS Mean = -1.5, 90% CI 2-sided [-5.7 to 2.8]
Statistical Analysis 18: Comparison: Group 2: Moxifloxacin 400 mg; Pre dose; Test type: Other; LS Mean = 2.3, 90% CI 2-sided [-1.0 to 5.6]
Statistical Analysis 19: Comparison: Group 2: Moxifloxacin 400 mg; 0.5 hr Post dose; Test type: Other; LS Mean = -1.6, 90% CI 2-sided [-5.4 to 2.2]
Statistical Analysis 20: Comparison: Group 2: Moxifloxacin 400 mg; 1 hr Post dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-3.8 to 4.3]
Statistical Analysis 21: Comparison: Group 2: Moxifloxacin 400 mg; 1.5 hr Post dose; Test type: Other; LS Mean = 4.0, 90% CI 2-sided [0.4 to 7.6]
Statistical Analysis 22: Comparison: Group 2: Moxifloxacin 400 mg; 2 hr Post dose; Test type: Other; LS Mean = 6.3, 90% CI 2-sided [2.7 to 10.0]
Statistical Analysis 23: Comparison: Group 2: Moxifloxacin 400 mg; 2.5 hr Post dose; Test type: Other; LS Mean = 6.4, 90% CI 2-sided [2.6 to 10.2]
Statistical Analysis 24: Comparison: Group 2: Moxifloxacin 400 mg; 3 hr Post dose; Test type: Other; LS Mean = 8.5, 90% CI 2-sided [5.0 to 12.0]
Statistical Analysis 25: Comparison: Group 2: Moxifloxacin 400 mg; 4 hr Post dose; Test type: Other; LS Mean = 10.1, 90% CI 2-sided [6.4 to 13.8]
Statistical Analysis 26: Comparison: Group 2: Moxifloxacin 400 mg; 5 hr Post dose; Test type: Other; LS Mean = 7.8, 90% CI 2-sided [4.1 to 11.6]
Statistical Analysis 27: Comparison: Group 2: Moxifloxacin 400 mg; 6 hr Post dose; Test type: Other; LS Mean = 7.8, 90% CI 2-sided [4.4 to 11.2]
Statistical Analysis 28: Comparison: Group 2: Moxifloxacin 400 mg; 7 hr Post dose; Test type: Other; LS Mean = 6.8, 90% CI 2-sided [3.4 to 10.2]
Statistical Analysis 29: Comparison: Group 2: Moxifloxacin 400 mg; 8 hr Post dose; Test type: Other; LS Mean = 4.5, 90% CI 2-sided [0.6 to 8.3]
Statistical Analysis 30: Comparison: Group 2: Moxifloxacin 400 mg; 9 hr Post dose; Test type: Other; LS Mean = 6.5, 90% CI 2-sided [3.1 to 10.0]
Statistical Analysis 31: Comparison: Group 2: Moxifloxacin 400 mg; 10 hr Post dose; Test type: Other; LS Mean = 6.6, 90% CI 2-sided [3.0 to 10.1]
Statistical Analysis 32: Comparison: Group 2: Moxifloxacin 400 mg; 12 hr Post dose; Test type: Other; LS Mean = 5.3, 90% CI 2-sided [1.8 to 8.8]
Statistical Analysis 33: Comparison: Group 2: Moxifloxacin 400 mg; 16 hr Post dose; Test type: Other; LS Mean = 7.2, 90% CI 2-sided [3.7 to 10.6]
Statistical Analysis 34: Comparison: Group 2: Moxifloxacin 400 mg; 24 hr Post dose; Test type: Other; LS Mean = 3.3, 90% CI 2-sided [-1.0 to 7.5]

6. Secondary Outcome: Placebo-corrected CHFB in QTcF Intervals After Administration of SC Setmelanotide or Oral Moxifloxacin at Day 16
Description: The CHFB in QTcF was analysed using an ANOVA including treatment, time and their interaction as main factors and structuring the residual matrix in order to account for the repeated measurement pattern of the data. HR was considered as covariate.
Time Frame: Baseline and Day 16: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Group 1: Setmelanotide 7 mg | Group 3: Moxifloxacin 400 mg
Number analyzed (Participants) | 21 | 25
msec
  Pre dose: number analyzed (Participants) | 21 | 24
  Pre dose | 4.5 (6.49) | -0.8 (8.30)
  0.5 hr Post dose | 1.0 (8.83) | -1.8 (5.93)
  1 hr Post dose | 1.6 (9.18) | -1.9 (7.49)
  1.5 hr Post dose: number analyzed (Participants) | 21 | 24
  1.5 hr Post dose | 0.3 (10.42) | 3.0 (7.05)
  2 hr Post dose | 2.2 (10.94) | 4.2 (7.53)
  2.5 hr Post dose | 2.7 (11.61) | 7.6 (8.45)
  3 hr Post dose | 4.3 (11.34) | 8.1 (8.19)
  4 hr Post dose: number analyzed (Participants) | 20 | 25
  4 hr Post dose | 3.6 (9.88) | 8.8 (6.37)
  5 hr Post dose: number analyzed (Participants) | 20 | 25
  5 hr Post dose | 4.7 (9.41) | 7.5 (8.97)
  6 hr Post dose: number analyzed (Participants) | 20 | 25
  6 hr Post dose | 2.8 (9.64) | 8.5 (6.18)
  7 hr Post dose | 1.5 (11.14) | 9.1 (7.29)
  8 hr Post dose: number analyzed (Participants) | 21 | 23
  8 hr Post dose | 2.8 (10.02) | 8.0 (5.73)
  9 hr Post dose: number analyzed (Participants) | 21 | 23
  9 hr Post dose | 6.1 (8.72) | 7.0 (7.33)
  10 hr Post dose | 6.5 (6.64) | 7.0 (9.93)
  12 hr Post dose: number analyzed (Participants) | 21 | 24
  12 hr Post dose | 5.8 (7.96) | 10.8 (9.14)
  16 hr Post dose: number analyzed (Participants) | 20 | 24
  16 hr Post dose | 1.4 (7.77) | 6.6 (8.51)
  24 hr Post dose: number analyzed (Participants) | 20 | 23
  24 hr Post dose | 1.0 (11.26) | 4.4 (10.57)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 7 mg; Pre dose; Test type: Other; LS Mean = 7.8, 90% CI 2-sided [3.7 to 11.8]
Statistical Analysis 2: Comparison: Group 1: Setmelanotide 7 mg; 0.5 hr Post dose; Test type: Other; LS Mean = 6.5, 90% CI 2-sided [3.3 to 9.8]
Statistical Analysis 3: Comparison: Group 1: Setmelanotide 7 mg; 1 hr Post dose; Test type: Other; LS Mean = 4.6, 90% CI 2-sided [0.6 to 8.6]
Statistical Analysis 4: Comparison: Group 1: Setmelanotide 7 mg; 1.5 hr Post dose; Test type: Other; LS Mean = 4.6, 90% CI 2-sided [0.6 to 8.6]
Statistical Analysis 5: Comparison: Group 1: Setmelanotide 7 mg; 2 hr Post dose; Test type: Other; LS Mean = 3.8, 90% CI 2-sided [-0.4 to 8.0]
Statistical Analysis 6: Comparison: Group 1: Setmelanotide 7 mg; 2.5 hr Post dose; Test type: Other; LS Mean = 6.1, 90% CI 2-sided [1.8 to 10.4]
Statistical Analysis 7: Comparison: Group 1: Setmelanotide 7 mg; 3 hr Post dose; Test type: Other; LS Mean = 5.7, 90% CI 2-sided [1.7 to 9.8]
Statistical Analysis 8: Comparison: Group 1: Setmelanotide 7 mg; 4 hr Post dose; Test type: Other; LS Mean = 6.2, 90% CI 2-sided [2.5 to 9.8]
Statistical Analysis 9: Comparison: Group 1: Setmelanotide 7 mg; 5 hr Post dose; Test type: Other; LS Mean = 5.7, 90% CI 2-sided [1.6 to 9.8]
Statistical Analysis 10: Comparison: Group 1: Setmelanotide 7 mg; 6 hr Post dose; Test type: Other; LS Mean = 4.8, 90% CI 2-sided [1.1 to 8.4]
Statistical Analysis 11: Comparison: Group 1: Setmelanotide 7 mg; 7 hr Post dose; Test type: Other; LS Mean = 3.0, 90% CI 2-sided [-0.9 to 7.0]
Statistical Analysis 12: Comparison: Group 1: Setmelanotide 7 mg; 8 hr Post dose; Test type: Other; LS Mean = 5.0, 90% CI 2-sided [1.3 to 8.8]
Statistical Analysis 13: Comparison: Group 1: Setmelanotide 7 mg; 9 hr Post dose; Test type: Other; LS Mean = 6.5, 90% CI 2-sided [2.5 to 10.6]
Statistical Analysis 14: Comparison: Group 1: Setmelanotide 7 mg; 10 hr Post dose; Test type: Other; LS Mean = 8.6, 90% CI 2-sided [4.8 to 12.3]
Statistical Analysis 15: Comparison: Group 1: Setmelanotide 7 mg; 12 hr Post dose; Test type: Other; LS Mean = 7.9, 90% CI 2-sided [4.4 to 11.4]
Statistical Analysis 16: Comparison: Group 1: Setmelanotide 7 mg; 16 hr Post dose; Test type: Other; LS Mean = 4.9, 90% CI 2-sided [0.9 to 8.9]
Statistical Analysis 17: Comparison: Group 1: Setmelanotide 7 mg; 24 hr Post dose; Test type: Other; LS Mean = 7.8, 90% CI 2-sided [3.6 to 12.0]
Statistical Analysis 18: Comparison: Group 3: Moxifloxacin 400 mg; Pre dose; Test type: Other; LS Mean = 2.1, 90% CI 2-sided [-1.8 to 6.0]
Statistical Analysis 19: Comparison: Group 3: Moxifloxacin 400 mg; 0.5 hr Post dose; Test type: Other; LS Mean = 3.1, 90% CI 2-sided [-0.0 to 6.2]
Statistical Analysis 20: Comparison: Group 3: Moxifloxacin 400 mg; 1 hr Post dose; Test type: Other; LS Mean = 1.9, 90% CI 2-sided [-1.9 to 5.7]
Statistical Analysis 21: Comparison: Group 3: Moxifloxacin 400 mg; 1.5 hr Post dose; Test type: Other; LS Mean = 6.5, 90% CI 2-sided [2.6 to 10.4]
Statistical Analysis 22: Comparison: Group 3: Moxifloxacin 400 mg; 2 hr Post dose; Test type: Other; LS Mean = 5.3, 90% CI 2-sided [1.3 to 9.3]
Statistical Analysis 23: Comparison: Group 3: Moxifloxacin 400 mg; 2.5 hr Post dose; Test type: Other; LS Mean = 11.1, 90% CI 2-sided [7.0 to 15.1]
Statistical Analysis 24: Comparison: Group 3: Moxifloxacin 400 mg; 3 hr Post dose; Test type: Other; LS Mean = 9.8, 90% CI 2-sided [5.9 to 13.6]
Statistical Analysis 25: Comparison: Group 3: Moxifloxacin 400 mg; 4 hr Post dose; Test type: Other; LS Mean = 10.7, 90% CI 2-sided [7.2 to 14.2]
Statistical Analysis 26: Comparison: Group 3: Moxifloxacin 400 mg; 5 hr Post dose; Test type: Other; LS Mean = 8.8, 90% CI 2-sided [4.9 to 12.7]
Statistical Analysis 27: Comparison: Group 3: Moxifloxacin 400 mg; 6 hr Post dose; Test type: Other; LS Mean = 11.0, 90% CI 2-sided [7.5 to 14.5]
Statistical Analysis 28: Comparison: Group 3: Moxifloxacin 400 mg; 7 hr Post dose; Test type: Other; LS Mean = 10.8, 90% CI 2-sided [7.1 to 14.6]
Statistical Analysis 29: Comparison: Group 3: Moxifloxacin 400 mg; 8 hr Post dose; Test type: Other; LS Mean = 11.3, 90% CI 2-sided [7.6 to 14.9]
Statistical Analysis 30: Comparison: Group 3: Moxifloxacin 400 mg; 9 hr Post dose; Test type: Other; LS Mean = 9.8, 90% CI 2-sided [5.9 to 13.7]
Statistical Analysis 31: Comparison: Group 3: Moxifloxacin 400 mg; 10 hr Post dose; Test type: Other; LS Mean = 10.5, 90% CI 2-sided [6.9 to 14.1]
Statistical Analysis 32: Comparison: Group 3: Moxifloxacin 400 mg; 12 hr Post dose; Test type: Other; LS Mean = 11.8, 90% CI 2-sided [8.4 to 15.2]
Statistical Analysis 33: Comparison: Group 3: Moxifloxacin 400 mg; 16 hr Post dose; Test type: Other; LS Mean = 9.4, 90% CI 2-sided [5.6 to 13.3]
Statistical Analysis 34: Comparison: Group 3: Moxifloxacin 400 mg; 24 hr Post dose; Test type: Other; LS Mean = 10.8, 90% CI 2-sided [6.8 to 14.9]

7. Secondary Outcome: Placebo-corrected CHFB in PR Intervals After Administration of SC Setmelanotide or Oral Moxifloxacin at Day 10
Description: The CHFB in PR was analyzed using an ANOVA including treatment, time and their interaction as main factors and structuring the residual matrix in order to account for the repeated measurement pattern of the data. HR was considered as covariate.
Time Frame: Baseline and Day 10: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Group 1: Setmelanotide 3 mg | Group 2: Moxifloxacin 400 mg
Number analyzed (Participants) | 23 | 23
msec
  Pre dose | -2.4 (6.12) | 3.1 (5.18)
  0.5 hr Post dose | -3.8 (8.93) | 3.4 (8.29)
  1 hr Post dose | -1.0 (6.22) | 3.5 (7.33)
  1.5 hr Post dose: number analyzed (Participants) | 23 | 21
  1.5 hr Post dose | -1.0 (6.24) | 3.7 (7.04)
  2 hr Post dose: number analyzed (Participants) | 23 | 21
  2 hr Post dose | -1.0 (6.98) | 3.3 (7.44)
  2.5 hr Post dose | -3.1 (4.92) | 1.5 (6.53)
  3 hr Post dose | -3.9 (7.81) | 2.6 (6.76)
  4 hr Post dose | -1.2 (5.78) | 1.6 (8.41)
  5 hr Post dose: number analyzed (Participants) | 23 | 22
  5 hr Post dose | -1.0 (6.61) | 0.5 (5.46)
  6 hr Post dose | -1.7 (5.87) | -0.2 (6.62)
  7 hr Post dose | -2.5 (4.88) | 0.3 (5.06)
  8 hr Post dose | -1.9 (7.06) | 0.3 (7.37)
  9 hr Post dose | -2.3 (6.03) | 0.5 (4.49)
  10 hr Post dose: number analyzed (Participants) | 23 | 22
  10 hr Post dose | -1.2 (7.06) | -0.8 (6.30)
  12 hr Post dose: number analyzed (Participants) | 23 | 22
  12 hr Post dose | -3.9 (7.83) | -2.1 (6.05)
  16 hr Post dose: number analyzed (Participants) | 22 | 22
  16 hr Post dose | -3.0 (7.02) | -0.0 (7.24)
  24 hr Post dose: number analyzed (Participants) | 21 | 22
  24 hr Post dose | -6.6 (8.39) | 1.2 (5.65)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 3 mg; Pre dose; Test type: Other; LS Mean = -5.3, 90% CI 2-sided [-8.4 to -2.2]
Statistical Analysis 2: Comparison: Group 2: Moxifloxacin 400 mg; 0.5 hr Post dose; Test type: Other; LS Mean = -2.7, 90% CI 2-sided [-5.9 to 0.5]
Statistical Analysis 3: Comparison: Group 1: Setmelanotide 3 mg; 1 hr Post dose; Test type: Other; LS Mean = -3.2, 90% CI 2-sided [-5.7 to -0.7]
Statistical Analysis 4: Comparison: Group 1: Setmelanotide 3 mg; 1.5 hr Post dose; Test type: Other; LS Mean = -0.9, 90% CI 2-sided [-3.7 to 1.9]
Statistical Analysis 5: Comparison: Group 1: Setmelanotide 3 mg; 2 hr Post dose; Test type: Other; LS Mean = -2.9, 90% CI 2-sided [-5.7 to -0.2]
Statistical Analysis 6: Comparison: Group 1: Setmelanotide 3 mg; 2.5 hr Post dose; Test type: Other; LS Mean = -4.0, 90% CI 2-sided [-6.5 to -1.5]
Statistical Analysis 7: Comparison: Group 1: Setmelanotide 3 mg; 3 hr Post dose; Test type: Other; LS Mean = -4.2, 90% CI 2-sided [-7.1 to -1.3]
Statistical Analysis 8: Comparison: Group 1: Setmelanotide 3 mg; 4 hr Post dose; Test type: Other; LS Mean = -4.1, 90% CI 2-sided [-7.4 to -0.8]
Statistical Analysis 9: Comparison: Group 1: Setmelanotide 3 mg; 5 hr Post dose; Test type: Other; LS Mean = -0.8, 90% CI 2-sided [-3.7 to 2.1]
Statistical Analysis 10: Comparison: Group 1: Setmelanotide 3 mg; 6 hr Post dose; Test type: Other; LS Mean = -3.3, 90% CI 2-sided [-6.3 to -0.4]
Statistical Analysis 11: Comparison: Group 1: Setmelanotide 3 mg; 7 hr Post dose; Test type: Other; LS Mean = -3.3, 90% CI 2-sided [-6.0 to -0.5]
Statistical Analysis 12: Comparison: Group 1: Setmelanotide 3 mg; 8 hr Post dose; Test type: Other; LS Mean = -1.6, 90% CI 2-sided [-4.7 to 1.5]
Statistical Analysis 13: Comparison: Group 1: Setmelanotide 3 mg; 9 hr Post dose; Test type: Other; LS Mean = -4.0, 90% CI 2-sided [-6.9 to -1.2]
Statistical Analysis 14: Comparison: Group 1: Setmelanotide 3 mg; 10 hr Post dose; Test type: Other; LS Mean = -4.3, 90% CI 2-sided [-7.6 to -1.0]
Statistical Analysis 15: Comparison: Group 1: Setmelanotide 3 mg; 12 hr Post dose; Test type: Other; LS Mean = -5.4, 90% CI 2-sided [-8.7 to -2.1]
Statistical Analysis 16: Comparison: Group 1: Setmelanotide 3 mg; 16 hr Post dose; Test type: Other; LS Mean = -4.1, 90% CI 2-sided [-7.4 to -0.8]
Statistical Analysis 17: Comparison: Group 1: Setmelanotide 3 mg; 24 hr Post dose; Test type: Other; LS Mean = -7.1, 90% CI 2-sided [-10.1 to -4.2]
Statistical Analysis 18: Comparison: Group 2: Moxifloxacin 400 mg; Pre dose; Test type: Other; LS Mean = 1.1, 90% CI 2-sided [-2.0 to 4.2]
Statistical Analysis 19: Comparison: Group 2: Moxifloxacin 400 mg; 0.5 hr Post dose; Test type: Other; LS Mean = 3.1, 90% CI 2-sided [-0.1 to 6.3]
Statistical Analysis 20: Comparison: Group 2: Moxifloxacin 400 mg; 1 hr Post dose; Test type: Other; LS Mean = 2.4, 90% CI 2-sided [-0.1 to 4.9]
Statistical Analysis 21: Comparison: Group 2: Moxifloxacin 400 mg; 1.5 hr Post dose; Test type: Other; LS Mean = 3.0, 90% CI 2-sided [0.2 to 5.8]
Statistical Analysis 22: Comparison: Group 2: Moxifloxacin 400 mg; 2 hr Post dose; Test type: Other; LS Mean = 1.8, 90% CI 2-sided [-1.0 to 4.6]
Statistical Analysis 23: Comparison: Group 2: Moxifloxacin 400 mg; 2.5 hr Post dose; Test type: Other; LS Mean = 0.6, 90% CI 2-sided [-1.9 to 3.1]
Statistical Analysis 24: Comparison: Group 2: Moxifloxacin 400 mg; 3 hr Post dose; Test type: Other; LS Mean = 1.9, 90% CI 2-sided [-1.0 to 4.8]
Statistical Analysis 25: Comparison: Group 2: Moxifloxacin 400 mg; 4 hr Post dose; Test type: Other; LS Mean = -0.3, 90% CI 2-sided [-3.5 to 3.0]
Statistical Analysis 26: Comparison: Group 2: Moxifloxacin 400 mg; 5 hr Post dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-2.6 to 3.2]
Statistical Analysis 27: Comparison: Group 2: Moxifloxacin 400 mg; 6 hr Post dose; Test type: Other; LS Mean = -1.9, 90% CI 2-sided [-4.8 to 1.1]
Statistical Analysis 28: Comparison: Group 2: Moxifloxacin 400 mg; 7 hr Post dose; Test type: Other; LS Mean = -1.1, 90% CI 2-sided [-3.8 to 1.7]
Statistical Analysis 29: Comparison: Group 2: Moxifloxacin 400 mg; 8 hr Post dose; Test type: Other; LS Mean = -0.5, 90% CI 2-sided [-3.6 to 2.6]
Statistical Analysis 30: Comparison: Group 2: Moxifloxacin 400 mg; 9 hr Post dose; Test type: Other; LS Mean = -2.7, 90% CI 2-sided [-5.6 to 0.2]
Statistical Analysis 31: Comparison: Group 2: Moxifloxacin 400 mg; 10 hr Post dose; Test type: Other; LS Mean = -3.5, 90% CI 2-sided [-6.8 to -0.2]
Statistical Analysis 32: Comparison: Group 2: Moxifloxacin 400 mg; 12 hr Post dose; Test type: Other; LS Mean = -3.3, 90% CI 2-sided [-6.6 to 0.1]
Statistical Analysis 33: Comparison: Group 2: Moxifloxacin 400 mg; 16 hr Post dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-3.0 to 3.6]
Statistical Analysis 34: Comparison: Group 2: Moxifloxacin 400 mg; 24 hr Post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-3.0 to 2.9]

8. Secondary Outcome: Placebo-corrected CHFB in PR Intervals After Administration of SC Setmelanotide or Oral Moxifloxacin at Day 16
Description: The CHFB in PR was analysed using an ANOVA including treatment, time and their interaction as main factors and structuring the residual matrix in order to account for the repeated measurement pattern of the data. HR was considered as covariate.
Time Frame: Baseline and Day 16: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Group 1: Setmelanotide 7 mg | Group 3: Moxifloxacin 400 mg
Number analyzed (Participants) | 21 | 25
msec
  Pre dose: number analyzed (Participants) | 21 | 24
  Pre dose | -3.5 (7.11) | 3.4 (11.46)
  0.5 hr Post dose | -4.5 (11.01) | 3.9 (9.88)
  1 hr Post dose | 0.4 (7.72) | 5.8 (10.90)
  1.5 hr Post dose: number analyzed (Participants) | 21 | 24
  1.5 hr Post dose | -2.3 (7.45) | 2.4 (9.42)
  2 hr Post dose | 0.1 (6.67) | 2.0 (8.17)
  2.5 hr Post dose | -0.9 (7.36) | 3.2 (7.46)
  3 hr Post dose | -2.2 (7.12) | 2.0 (8.00)
  4 hr Post dose: number analyzed (Participants) | 20 | 25
  4 hr Post dose | -1.3 (6.34) | 1.3 (9.51)
  5 hr Post dose: number analyzed (Participants) | 20 | 22
  5 hr Post dose | -2.6 (6.70) | 1.2 (9.99)
  6 hr Post dose: number analyzed (Participants) | 20 | 25
  6 hr Post dose | -1.7 (7.99) | 0.7 (8.87)
  7 hr Post dose | -3.7 (5.65) | -1.1 (9.29)
  8 hr Post dose: number analyzed (Participants) | 21 | 23
  8 hr Post dose | -3.1 (5.97) | 0.8 (8.52)
  9 hr Post dose: number analyzed (Participants) | 21 | 23
  9 hr Post dose | -3.4 (5.08) | 0.4 (7.66)
  10 hr Post dose | -1.4 (6.36) | 1.1 (7.80)
  12 hr Post dose: number analyzed (Participants) | 21 | 24
  12 hr Post dose | -1.9 (5.77) | 0.8 (7.27)
  16 hr Post dose: number analyzed (Participants) | 20 | 24
  16 hr Post dose | -4.9 (6.64) | 0.9 (8.78)
  24 hr Post dose: number analyzed (Participants) | 20 | 23
  24 hr Post dose | -8.4 (9.21) | 2.5 (7.28)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 7 mg; Pre dose; Test type: Other; LS Mean = -6.6, 90% CI 2-sided [-10.3 to -3.0]
Statistical Analysis 2: Comparison: Group 1: Setmelanotide 7 mg; 0.5 hr Post dose; Test type: Other; LS Mean = -7.3, 90% CI 2-sided [-10.5 to -4.0]
Statistical Analysis 3: Comparison: Group 1: Setmelanotide 7 mg; 1 hr Post dose; Test type: Other; LS Mean = -5.0, 90% CI 2-sided [-8.8 to -1.2]
Statistical Analysis 4: Comparison: Group 1: Setmelanotide 7 mg; 1.5 hr Post dose; Test type: Other; LS Mean = -5.0, 90% CI 2-sided [-8.4 to -1.6]
Statistical Analysis 5: Comparison: Group 1: Setmelanotide 7 mg; 2 hr Post dose; Test type: Other; LS Mean = -3.5, 90% CI 2-sided [-6.6 to -0.3]
Statistical Analysis 6: Comparison: Group 1: Setmelanotide 7 mg; 2.5 hr Post dose; Test type: Other; LS Mean = -2.9, 90% CI 2-sided [-6.1 to 0.3]
Statistical Analysis 7: Comparison: Group 1: Setmelanotide 7 mg; 3 hr Post dose; Test type: Other; LS Mean = -4.6, 90% CI 2-sided [-7.7 to -1.5]
Statistical Analysis 8: Comparison: Group 1: Setmelanotide 7 mg; 4 hr Post dose; Test type: Other; LS Mean = -7.1, 90% CI 2-sided [-10.3 to -3.8]
Statistical Analysis 9: Comparison: Group 1: Setmelanotide 7 mg; 5 hr Post dose; Test type: Other; LS Mean = -3.2, 90% CI 2-sided [-6.9 to 0.6]
Statistical Analysis 10: Comparison: Group 1: Setmelanotide 7 mg; 6 hr Post dose; Test type: Other; LS Mean = -4.2, 90% CI 2-sided [-7.8 to -0.6]
Statistical Analysis 11: Comparison: Group 1: Setmelanotide 7 mg; 7 hr Post dose; Test type: Other; LS Mean = -4.8, 90% CI 2-sided [-8.1 to -1.6]
Statistical Analysis 12: Comparison: Group 1: Setmelanotide 7 mg; 8 hr Post dose; Test type: Other; LS Mean = -4.4, 90% CI 2-sided [-7.8 to -1.1]
Statistical Analysis 13: Comparison: Group 1: Setmelanotide 7 mg; 9 hr Post dose; Test type: Other; LS Mean = -5.9, 90% CI 2-sided [-9.3 to -2.6]
Statistical Analysis 14: Comparison: Group 1: Setmelanotide 7 mg; 10 hr Post dose; Test type: Other; LS Mean = -4.4, 90% CI 2-sided [-7.8 to -1.1]
Statistical Analysis 15: Comparison: Group 1: Setmelanotide 7 mg; 12 hr Post dose; Test type: Other; LS Mean = -4.2, 90% CI 2-sided [-7.3 to -1.1]
Statistical Analysis 16: Comparison: Group 1: Setmelanotide 7 mg; 16 hr Post dose; Test type: Other; LS Mean = -5.8, 90% CI 2-sided [-9.7 to -2.0]
Statistical Analysis 17: Comparison: Group 1: Setmelanotide 7 mg; 24 hr Post dose; Test type: Other; LS Mean = -8.2, 90% CI 2-sided [-12.5 to -3.8]
Statistical Analysis 18: Comparison: Group 3: Moxifloxacin 400 mg; Pre dose; Test type: Other; LS Mean = 2.4, 90% CI 2-sided [-1.2 to 5.9]
Statistical Analysis 19: Comparison: Group 3: Moxifloxacin 400 mg; 0.5 hr Post dose; Test type: Other; LS Mean = -1.4, 90% CI 2-sided [-4.5 to 1.8]
Statistical Analysis 20: Comparison: Group 3: Moxifloxacin 400 mg; 1 hr Post dose; Test type: Other; LS Mean = -0.4, 90% CI 2-sided [-4.0 to 3.3]
Statistical Analysis 21: Comparison: Group 3: Moxifloxacin 400 mg; 1.5 hr Post dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-3.0 to 3.6]
Statistical Analysis 22: Comparison: Group 3: Moxifloxacin 400 mg; 2 hr Post dose; Test type: Other; LS Mean = -1.0, 90% CI 2-sided [-4.0 to 2.0]
Statistical Analysis 23: Comparison: Group 3: Moxifloxacin 400 mg; 2.5 hr Post dose; Test type: Other; LS Mean = 0.5, 90% CI 2-sided [-2.6 to 3.6]
Statistical Analysis 24: Comparison: Group 3: Moxifloxacin 400 mg; 3 hr Post dose; Test type: Other; LS Mean = -0.7, 90% CI 2-sided [-3.7 to 2.3]
Statistical Analysis 25: Comparison: Group 3: Moxifloxacin 400 mg; 4 hr Post dose; Test type: Other; LS Mean = -2.3, 90% CI 2-sided [-5.4 to 0.9]
Statistical Analysis 26: Comparison: Group 3: Moxifloxacin 400 mg; 5 hr Post dose; Test type: Other; LS Mean = 1.1, 90% CI 2-sided [-2.5 to 4.6]
Statistical Analysis 27: Comparison: Group 3: Moxifloxacin 400 mg; 6 hr Post dose; Test type: Other; LS Mean = -0.7, 90% CI 2-sided [-4.1 to 2.8]
Statistical Analysis 28: Comparison: Group 3: Moxifloxacin 400 mg; 7 hr Post dose; Test type: Other; LS Mean = -1.9, 90% CI 2-sided [-5.0 to 1.3]
Statistical Analysis 29: Comparison: Group 3: Moxifloxacin 400 mg; 8 hr Post dose; Test type: Other; LS Mean = -0.5, 90% CI 2-sided [-3.7 to 2.8]
Statistical Analysis 30: Comparison: Group 3: Moxifloxacin 400 mg; 9 hr Post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-3.4 to 3.1]
Statistical Analysis 31: Comparison: Group 3: Moxifloxacin 400 mg; 10 hr Post dose; Test type: Other; LS Mean = 0.4, 90% CI 2-sided [-2.8 to 3.7]
Statistical Analysis 32: Comparison: Group 3: Moxifloxacin 400 mg; 12 hr Post dose; Test type: Other; LS Mean = 0.1, 90% CI 2-sided [-2.9 to 3.1]
Statistical Analysis 33: Comparison: Group 3: Moxifloxacin 400 mg; 16 hr Post dose; Test type: Other; LS Mean = 0.6, 90% CI 2-sided [-3.1 to 4.3]
Statistical Analysis 34: Comparison: Group 3: Moxifloxacin 400 mg; 24 hr Post dose; Test type: Other; LS Mean = 1.7, 90% CI 2-sided [-2.5 to 5.9]

9. Secondary Outcome: Placebo-corrected CHFB in QRS Intervals After Administration of SC Setmelanotide or Oral Moxifloxacin at Day 10
Description: The CHFB in QRS was analysed using an ANOVA including treatment, time and their interaction as main factors and structuring the residual matrix in order to account for the repeated measurement pattern of the data. HR was considered as covariate.
Time Frame: Baseline and Day 10: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Group 1: Setmelanotide 3 mg | Group 2: Moxifloxacin 400 mg
Number analyzed (Participants) | 23 | 23
msec
  Pre dose | -0.2 (4.90) | 0.9 (3.42)
  0.5 hr Post dose | 0.0 (3.85) | 0.6 (6.31)
  1 hr Post dose | 0.5 (5.21) | 0.8 (3.38)
  1.5 hr Post dose: number analyzed (Participants) | 23 | 21
  1.5 hr Post dose | -0.6 (3.69) | -0.2 (3.06)
  2 hr Post dose: number analyzed (Participants) | 23 | 21
  2 hr Post dose | 0.2 (4.04) | 0.1 (3.37)
  2.5 hr Post dose | 0.2 (4.41) | 0.5 (4.70)
  3 hr Post dose | 0.7 (4.31) | 0.4 (3.60)
  4 hr Post dose | 0.6 (3.95) | -0.7 (3.94)
  5 hr Post dose: number analyzed (Participants) | 23 | 22
  5 hr Post dose | 0.5 (3.82) | 1.0 (3.88)
  6 hr Post dose | 0.4 (4.71) | -0.4 (3.92)
  7 hr Post dose | 0.9 (5.30) | 0.1 (3.66)
  8 hr Post dose | 0.2 (4.23) | 1.1 (3.85)
  9 hr Post dose: number analyzed (Participants) | 23 | 22
  9 hr Post dose | -0.2 (4.19) | -0.1 (2.93)
  10 hr Post dose: number analyzed (Participants) | 23 | 22
  10 hr Post dose | 1.6 (4.23) | 0.2 (3.95)
  12 hr Post dose: number analyzed (Participants) | 23 | 22
  12 hr Post dose | 0.8 (5.08) | 1.9 (4.10)
  16 hr Post dose: number analyzed (Participants) | 22 | 22
  16 hr Post dose | 1.0 (4.77) | 1.5 (3.97)
  24 hr Post dose: number analyzed (Participants) | 21 | 22
  24 hr Post dose | -0.3 (5.38) | 1.6 (4.53)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 3 mg; Pre dose; Test type: Other; LS Mean = -0.7, 90% CI 2-sided [-2.6 to 1.2]
Statistical Analysis 2: Comparison: Group 1: Setmelanotide 3 mg; 0.5 hr post dose; Test type: Other; LS Mean = -0.9, 90% CI 2-sided [-2.6 to 0.7]
Statistical Analysis 3: Comparison: Group 1: Setmelanotide 3 mg; 1 hr post dose; Test type: Other; LS Mean = 0.6, 90% CI 2-sided [-1.1 to 2.3]
Statistical Analysis 4: Comparison: Group 1: Setmelanotide 3 mg; 1.5 hr post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-1.5 to 1.3]
Statistical Analysis 5: Comparison: Group 1: Setmelanotide 3 mg; 2 hr post dose; Test type: Other; LS Mean = 0.8, 90% CI 2-sided [-0.8 to 2.4]
Statistical Analysis 6: Comparison: Group 1: Setmelanotide 3 mg; 2.5 hr post dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-1.0 to 2.4]
Statistical Analysis 7: Comparison: Group 1: Setmelanotide 3 mg; 3 hr post dose; Test type: Other; LS Mean = 0.2, 90% CI 2-sided [-1.6 to 2.0]
Statistical Analysis 8: Comparison: Group 1: Setmelanotide 3 mg; 4 hr post dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-0.9 to 2.3]
Statistical Analysis 9: Comparison: Group 1: Setmelanotide 3 mg; 5 hr post dose; Test type: Other; LS Mean = 0.5, 90% CI 2-sided [-1.2 to 2.1]
Statistical Analysis 10: Comparison: Group 1: Setmelanotide 3 mg; 6 hr post dose; Test type: Other; LS Mean = 0.9, 90% CI 2-sided [-0.7 to 2.4]
Statistical Analysis 11: Comparison: Group 1: Setmelanotide 3 mg; 7 hr post dose; Test type: Other; LS Mean = 0.9, 90% CI 2-sided [-0.6 to 2.4]
Statistical Analysis 12: Comparison: Group 1: Setmelanotide 3 mg; 8 hr post dose; Test type: Other; LS Mean = 0.6, 90% CI 2-sided [-1.0 to 2.2]
Statistical Analysis 13: Comparison: Group 1: Setmelanotide 3 mg; 9 hr post dose; Test type: Other; LS Mean = -0.2, 90% CI 2-sided [-1.6 to 1.3]
Statistical Analysis 14: Comparison: Group 1: Setmelanotide 3 mg; 10 hr post dose; Test type: Other; LS Mean = 0.0, 90% CI 2-sided [-1.5 to 1.6]
Statistical Analysis 15: Comparison: Group 1: Setmelanotide 3 mg; 12 hr post dose; Test type: Other; LS Mean = 1.4, 90% CI 2-sided [-0.2 to 3.0]
Statistical Analysis 16: Comparison: Group 1: Setmelanotide 3 mg; 16 hr post dose; Test type: Other; LS Mean = 1.5, 90% CI 2-sided [-0.3 to 3.4]
Statistical Analysis 17: Comparison: Group 1: Setmelanotide 3 mg; 24 hr post dose; Test type: Other; LS Mean = -0.2, 90% CI 2-sided [-2.1 to 1.6]
Statistical Analysis 18: Comparison: Group 2: Moxifloxacin 400 mg; Pre dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-1.2 to 2.6]
Statistical Analysis 19: Comparison: Group 2: Moxifloxacin 400 mg; 0.5 hr post dose; Test type: Other; LS Mean = -0.3, 90% CI 2-sided [-1.9 to 1.4]
Statistical Analysis 20: Comparison: Group 2: Moxifloxacin 400 mg; 1 hr post dose; Test type: Other; LS Mean = 0.5, 90% CI 2-sided [-1.2 to 2.2]
Statistical Analysis 21: Comparison: Group 2: Moxifloxacin 400 mg; 1.5 hr post dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-0.7 to 2.1]
Statistical Analysis 22: Comparison: Group 2: Moxifloxacin 400 mg; 2 hr post dose; Test type: Other; LS Mean = 0.6, 90% CI 2-sided [-1.1 to 2.2]
Statistical Analysis 23: Comparison: Group 2: Moxifloxacin 400 mg; 2.5 hr post dose; Test type: Other; LS Mean = 0.8, 90% CI 2-sided [-0.9 to 2.5]
Statistical Analysis 24: Comparison: Group 2: Moxifloxacin 400 mg; 3 hr post dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-1.5 to 2.1]
Statistical Analysis 25: Comparison: Group 2: Moxifloxacin 400 mg; 4 hr post dose; Test type: Other; LS Mean = -0.5, 90% CI 2-sided [-2.1 to 1.1]
Statistical Analysis 26: Comparison: Group 2: Moxifloxacin 400 mg; 5 hr post dose; Test type: Other; LS Mean = 0.2, 90% CI 2-sided [-1.5 to 1.9]
Statistical Analysis 27: Comparison: Group 2: Moxifloxacin 400 mg; 6 hr post dose; Test type: Other; LS Mean = -0.2, 90% CI 2-sided [-1.7 to 1.4]
Statistical Analysis 28: Comparison: Group 2: Moxifloxacin 400 mg; 7 hr post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-1.6 to 1.4]
Statistical Analysis 29: Comparison: Group 2: Moxifloxacin 400 mg; 8 hr post dose; Test type: Other; LS Mean = 0.8, 90% CI 2-sided [-0.7 to 2.4]
Statistical Analysis 30: Comparison: Group 2: Moxifloxacin 400 mg; 9 hr post dose; Test type: Other; LS Mean = -0.2, 90% CI 2-sided [-1.6 to 1.3]
Statistical Analysis 31: Comparison: Group 2: Moxifloxacin 400 mg; 10 hr post dose; Test type: Other; LS Mean = 0.1, 90% CI 2-sided [-1.4 to 1.6]
Statistical Analysis 32: Comparison: Group 2: Moxifloxacin 400 mg; 12 hr post dose; Test type: Other; LS Mean = 1.5, 90% CI 2-sided [-0.1 to 3.1]
Statistical Analysis 33: Comparison: Group 2: Moxifloxacin 400 mg; 16 hr post dose; Test type: Other; LS Mean = 1.2, 90% CI 2-sided [-0.7 to 3.0]
Statistical Analysis 34: Comparison: Group 2: Moxifloxacin 400 mg; 24 hr post dose; Test type: Other; LS Mean = 1.5, 90% CI 2-sided [-0.3 to 3.4]

10. Secondary Outcome: Placebo-corrected CHFB in QRS Intervals After Administration of SC Setmelanotide or Oral Moxifloxacin at Day 16
Description: The CHFB in QRS was analyzed using an ANOVA including treatment, time and their interaction as main factors and structuring the residual matrix in order to account for the repeated measurement pattern of the data. HR was considered as covariate.
Time Frame: Baseline and Day 16: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Group 1: Setmelanotide 7 mg | Group 3: Moxifloxacin 400 mg
Number analyzed (Participants) | 21 | 25
msec
  Pre dose: number analyzed (Participants) | 21 | 24
  Pre dose | 1.0 (4.11) | -0.8 (3.90)
  0.5 hr Post dose | 0.5 (3.57) | 0.2 (3.90)
  1 hr Post dose | 0.9 (3.20) | -1.0 (6.86)
  1.5 hr Post dose: number analyzed (Participants) | 21 | 24
  1.5 hr Post dose | -0.8 (3.06) | -0.4 (3.65)
  2 hr Post dose | -0.2 (3.97) | 0.3 (3.41)
  2.5 hr Post dose | 1.1 (2.95) | -0.2 (4.20)
  3 hr Post dose | 0.5 (2.91) | 1.0 (3.69)
  4 hr Post dose: number analyzed (Participants) | 20 | 25
  4 hr Post dose | 0.7 (4.35) | 0.5 (2.93)
  5 hr Post dose: number analyzed (Participants) | 20 | 25
  5 hr Post dose | -0.2 (4.31) | -1.4 (5.54)
  6 hr Post dose: number analyzed (Participants) | 20 | 25
  6 hr Post dose | -0.2 (4.63) | 0.3 (2.99)
  7 hr Post dose | 1.5 (4.92) | 0.7 (4.10)
  8 hr Post dose: number analyzed (Participants) | 21 | 23
  8 hr Post dose | -0.2 (4.03) | 0.7 (2.77)
  9 hr Post dose: number analyzed (Participants) | 21 | 23
  9 hr Post dose | 0.2 (4.13) | -0.4 (3.15)
  10 hr Post dose | 1.2 (3.19) | -1.2 (2.73)
  12 hr Post dose: number analyzed (Participants) | 21 | 24
  12 hr Post dose | 1.4 (5.13) | -0.2 (4.74)
  16 hr Post dose: number analyzed (Participants) | 20 | 24
  16 hr Post dose | 1.1 (2.90) | -0.7 (4.75)
  24 hr Post dose: number analyzed (Participants) | 20 | 23
  24 hr Post dose | 1.3 (4.68) | 0.5 (3.69)
Statistical Analysis 1: Comparison: Group 1: Setmelanotide 7 mg; Pre dose; Test type: Other; LS Mean = 0.8, 90% CI 2-sided [-1.3 to 2.9]
Statistical Analysis 2: Comparison: Group 1: Setmelanotide 7 mg; 0.5 hr post dose; Test type: Other; LS Mean = -0.3, 90% CI 2-sided [-1.8 to 1.2]
Statistical Analysis 3: Comparison: Group 1: Setmelanotide 7 mg; 1 hr post dose; Test type: Other; LS Mean = 1.2, 90% CI 2-sided [-1.4 to 3.8]
Statistical Analysis 4: Comparison: Group 1: Setmelanotide 7 mg; 1.5 hr post dose; Test type: Other; LS Mean = -0.0, 90% CI 2-sided [-1.8 to 1.8]
Statistical Analysis 5: Comparison: Group 1: Setmelanotide 7 mg; 2 hr post dose; Test type: Other; LS Mean = -1.4, 90% CI 2-sided [-3.0 to 0.3]
Statistical Analysis 6: Comparison: Group 1: Setmelanotide 7 mg; 2.5 hr post dose; Test type: Other; LS Mean = 1.6, 90% CI 2-sided [-0.0 to 3.1]
Statistical Analysis 7: Comparison: Group 1: Setmelanotide 7 mg; 3 hr post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-1.7 to 1.5]
Statistical Analysis 8: Comparison: Group 1: Setmelanotide 7 mg; 4 hr post dose; Test type: Other; LS Mean = 1.3, 90% CI 2-sided [-0.3 to 2.9]
Statistical Analysis 9: Comparison: Group 1: Setmelanotide 7 mg; 5 hr post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-2.2 to 2.0]
Statistical Analysis 10: Comparison: Group 1: Setmelanotide 7 mg; 6 hr post dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-0.8 to 2.3]
Statistical Analysis 11: Comparison: Group 1: Setmelanotide 7 mg; 7 hr post dose; Test type: Other; LS Mean = 0.9, 90% CI 2-sided [-0.8 to 2.7]
Statistical Analysis 12: Comparison: Group 1: Setmelanotide 7 mg; 8 hr post dose; Test type: Other; LS Mean = 1.0, 90% CI 2-sided [-0.3 to 2.4]
Statistical Analysis 13: Comparison: Group 1: Setmelanotide 7 mg; 9 hr post dose; Test type: Other; LS Mean = 1.1, 90% CI 2-sided [-0.7 to 2.9]
Statistical Analysis 14: Comparison: Group 1: Setmelanotide 7 mg; 10 hr post dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-1.4 to 1.9]
Statistical Analysis 15: Comparison: Group 1: Setmelanotide 7 mg; 12 hr post dose; Test type: Other; LS Mean = 1.3, 90% CI 2-sided [-0.6 to 3.2]
Statistical Analysis 16: Comparison: Group 1: Setmelanotide 7 mg; 16 hr post dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-1.0 to 2.4]
Statistical Analysis 17: Comparison: Group 1: Setmelanotide 7 mg; 24 hr post dose; Test type: Other; LS Mean = 1.6, 90% CI 2-sided [-1.0 to 4.2]
Statistical Analysis 18: Comparison: Group 3: Moxifloxacin 400 mg; Pre dose; Test type: Other; LS Mean = -0.3, 90% CI 2-sided [-2.3 to 1.7]
Statistical Analysis 19: Comparison: Group 3: Moxifloxacin 400 mg; 0.5 hr post dose; Test type: Other; LS Mean = -0.1, 90% CI 2-sided [-1.6 to 1.3]
Statistical Analysis 20: Comparison: Group 3: Moxifloxacin 400 mg; 1 hr post dose; Test type: Other; LS Mean = -1.3, 90% CI 2-sided [-3.8 to 1.2]
Statistical Analysis 21: Comparison: Group 1: Setmelanotide 7 mg; 1.5 hr post dose; Test type: Other; LS Mean = 0.1, 90% CI 2-sided [-1.7 to 1.8]
Statistical Analysis 22: Comparison: Group 3: Moxifloxacin 400 mg; 2 hr post dose; Test type: Other; LS Mean = -1.1, 90% CI 2-sided [-2.7 to 0.5]
Statistical Analysis 23: Comparison: Group 3: Moxifloxacin 400 mg; 2.5 hr post dose; Test type: Other; LS Mean = 0.7, 90% CI 2-sided [-0.8 to 2.3]
Statistical Analysis 24: Comparison: Group 3: Moxifloxacin 400 mg; 3 hr post dose; Test type: Other; LS Mean = 0.2, 90% CI 2-sided [-1.3 to 1.8]
Statistical Analysis 25: Comparison: Group 3: Moxifloxacin 400 mg; 4 hr post dose; Test type: Other; LS Mean = 0.3, 90% CI 2-sided [-1.2 to 1.9]
Statistical Analysis 26: Comparison: Group 1: Setmelanotide 7 mg; 5 hr post dose; Test type: Other; LS Mean = -1.5, 90% CI 2-sided [-3.5 to 0.5]
Statistical Analysis 27: Comparison: Group 3: Moxifloxacin 400 mg; 6 hr post dose; Test type: Other; LS Mean = 0.9, 90% CI 2-sided [-0.6 to 2.3]
Statistical Analysis 28: Comparison: Group 3: Moxifloxacin 400 mg; 7 hr post dose; Test type: Other; LS Mean = 0.4, 90% CI 2-sided [-1.3 to 2.1]
Statistical Analysis 29: Comparison: Group 3: Moxifloxacin 400 mg; 8 hr post dose; Test type: Other; LS Mean = 1.3, 90% CI 2-sided [-0.0 to 2.6]
Statistical Analysis 30: Comparison: Group 3: Moxifloxacin 400 mg; 9 hr post dose; Test type: Other; LS Mean = 0.4, 90% CI 2-sided [-1.3 to 2.2]
Statistical Analysis 31: Comparison: Group 3: Moxifloxacin 400 mg; 10 hr post dose; Test type: Other; LS Mean = -1.1, 90% CI 2-sided [-2.7 to 0.5]
Statistical Analysis 32: Comparison: Group 3: Moxifloxacin 400 mg; 12 hr post dose; Test type: Other; LS Mean = -0.3, 90% CI 2-sided [-2.1 to 1.5]
Statistical Analysis 33: Comparison: Group 3: Moxifloxacin 400 mg; 16 hr post dose; Test type: Other; LS Mean = -0.2, 90% CI 2-sided [-1.9 to 1.4]
Statistical Analysis 34: Comparison: Group 3: Moxifloxacin 400 mg; 24 hr post dose; Test type: Other; LS Mean = 2.3, 90% CI 2-sided [-0.2 to 4.9]

11. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Abnormal Value in HR Intervals After Administration of SC Setmelanotide
Description: A treatment-emergent abnormality/finding was defined as any abnormality/finding not already reported on any of the ECGs collected before the administration. Abnormal findings included:
  HR (<40 beats/min, HR>120 beats/min and Relative CHFB >25%) Relative CHFB = 100*(Value-Baseline)/Baseline
Time Frame: Day 10 (for setmelanotide 3 mg) and Day 16 (for setmelanotide 7mg)
Population: ECG population with available data was analyzed. ECG data was collected on Days 10 and 16, where participants received setmelanotide 3 mg and 7 mg respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Setmelanotide 3 mg | Group 1: Setmelanotide 7 mg
Number analyzed (Participants) | 23 | 21
Participants
  HR<40 beats/min | 0 | 0
  HR>120 beats/min | 0 | 0
  Relative CHFB in HR>25% | 4 | 9

12. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Abnormal Value in PR Intervals After Administration of SC Setmelanotide
Description: A treatment-emergent abnormality/finding was defined as any abnormality/finding not already reported on any of the ECGs collected before the administration. Abnormal findings included:
  PR (>220 msec, Relative CHFB >25%); Relative CHFB = 100*(Value-Baseline)/Baseline
Time Frame: Day 10 (for setmelanotide 3 mg) and Day 16 (for setmelanotide 7mg)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Setmelanotide 3 mg | Group 1: Setmelanotide 7 mg
Number analyzed (Participants) | 23 | 21
Participants
  PR>220 msec | 0 | 0
  Relative CHFB in PR>25% | 0 | 0

13. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Abnormal Value in QRS Intervals After Administration of SC Setmelanotide
Description: A treatment-emergent abnormality/finding was defined as any abnormality/finding not already reported on any of the ECGs collected before the administration. Abnormal findings included:
  QRS ( >120 msec, Relative CHFB >25%); Relative CHFB = 100*(Value-Baseline)/Baseline
Time Frame: Day 10 (for setmelanotide 3 mg) and Day 16 (for setmelanotide 7mg)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Setmelanotide 3 mg | Group 1: Setmelanotide 7 mg
Number analyzed (Participants) | 23 | 21
Participants
  QRS>120 msec | 0 | 0
  Relative CHFB in QRS>25% | 0 | 0

14. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Abnormal Value in QTcF Intervals After Administration of SC Setmelanotide
Description: A treatment-emergent abnormality/finding was defined as any abnormality/finding not already reported on any of the ECGs collected before the administration. Abnormal findings included:
  QTcF (450<QTc<=480 msec, 480<QTc<=500 msec, QTc>500 msec, 30<CHFB in QTc<=60 msec, CHFB in >60 msec)
Time Frame: Day 10 (for setmelanotide 3 mg) and Day 16 (for setmelanotide 7mg)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Setmelanotide 3 mg | Group 1: Setmelanotide 7 mg
Number analyzed (Participants) | 23 | 21
Participants
  450<QTc<=480 msec | 0 | 0
  480<QTc<=500 msec | 0 | 0
  QTc>500 msec | 0 | 0
  30<CHFB in QTc<=60 msec | 0 | 0
  CHFB in QTc>60 msec | 0 | 0

15. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Abnormal Finding in T-wave Morphology and U-wave Presence After Administration of SC Setmelanotide
Description: A treatment-emergent abnormality/finding will be defined as any abnormality/finding not already reported on any of the ECGs collected before the administration.
  Abnormal findings included : QTcF Increase From Baseline, > 30 msec And < 60 msec
Time Frame: Day 10 (for setmelanotide 3 mg) and Day 16 (for setmelanotide 7mg)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Setmelanotide 3 mg | Group 1: Setmelanotide 7 mg
Number analyzed (Participants) | 23 | 23
Participants | 1 | 1

16. Secondary Outcome: Moxifloxacin Concentration-related CHFB in QTcF at Day 10
Description: Continuous 12-lead digital ECG recording was performed on Baseline and Day 10. ECG analysts were blinded to the treatment, timepoint and participant. CHFB in QTcF was calculated at each timepoint.
Time Frame: Baseline and Day 10: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: PK/QTc Population was analyzed. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Group 2: Moxifloxacin 400 mg
Number analyzed (Participants) | 23
msec
  Pre dose | 1.5 (7.76)
  0.5 hr Post dose | -5.3 (8.75)
  1 hr Post dose | -3.7 (9.39)
  1.5 hr Post dose: number analyzed (Participants) | 21
  1.5 hr Post dose | 0.9 (8.56)
  2 hr Post dose: number analyzed (Participants) | 21
  2 hr Post dose | 2.0 (8.74)
  2.5 hr Post dose | 4.9 (8.75)
  3 hr Post dose | 4.9 (7.39)
  4 hr Post dose | 6.3 (8.63)
  5 hr Post dose: number analyzed (Participants) | 22
  5 hr Post dose | 8.1 (8.42)
  6 hr Post dose | 6.0 (6.61)
  7 hr Post dose | 5.1 (8.39)
  8 hr Post dose | 4.4 (8.18)
  9 hr Post dose: number analyzed (Participants) | 22
  9 hr Post dose | 5.0 (10.47)
  10 hr Post dose: number analyzed (Participants) | 22
  10 hr Post dose | 6.2 (6.85)
  12 hr Post dose: number analyzed (Participants) | 22
  12 hr Post dose | 8.7 (4.84)
  16 hr Post dose: number analyzed (Participants) | 22
  16 hr Post dose | 5.9 (8.09)
  24 hr Post dose: number analyzed (Participants) | 22
  24 hr Post dose | 6.6 (8.00)

17. Secondary Outcome: Moxifloxacin Concentration-related CHFB in QTcF at Day 16
Description: Continuous 12-lead digital ECG recording was performed on Baseline and Day 16. ECG analysts were blinded to the treatment, timepoint and participant. CHFB in QTcF was calculated at each timepoint.
Time Frame: Baseline and Day 16: Pre dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10,12, 16, 24 hrs postdose
Population: PK/QTc Population was analyzed. Participants with available data were reported.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Group 3: Moxifloxacin 400 mg
Number analyzed (Participants) | 25
msec
  Pre dose: number analyzed (Participants) | 24
  Pre dose | -0.8 (8.30)
  0.5 hr Post dose | -1.8 (5.93)
  1 hr Post dose | -1.9 (7.49)
  1.5 hr Post dose: number analyzed (Participants) | 24
  1.5 hr Post dose | 3.0 (7.05)
  2 hr Post dose | 4.2 (7.53)
  2.5 hr Post dose | 7.6 (8.45)
  3 hr Post dose | 8.1 (8.19)
  4 hr Post dose | 8.8 (6.37)
  5 hr Post dose | 7.5 (8.97)
  6 hr Post dose | 8.5 (6.18)
  7 hr Post dose | 9.1 (7.29)
  8 hr Post dose: number analyzed (Participants) | 23
  8 hr Post dose | 8.0 (5.73)
  9 hr Post dose: number analyzed (Participants) | 23
  9 hr Post dose | 7.0 (7.33)
  10 hr Post dose | 7.0 (9.93)
  12 hr Post dose: number analyzed (Participants) | 24
  12 hr Post dose | 10.8 (9.14)
  16 hr Post dose: number analyzed (Participants) | 24
  16 hr Post dose | 6.6 (8.51)
  24 hr Post dose: number analyzed (Participants) | 23
  24 hr Post dose | 4.4 (10.57)

ADVERSE EVENTS:
Time Frame: From first dose up to Day 23
Description: The Safety population included all participants who received at least one dose of study drug.
Groups:
- Group 1: Setmelanotide 2 mg: Participants received once daily setmelanotide 2 mg from Days 1 to 7, via SC injection.
- Group 1: Setmelanotide 5 mg: Participants received once daily setmelanotide 5 mg from Days 11 to 13, via SC injection.
- Group 2: Placebo: Participants received once daily Placebo from Days 1 to 16, via SC injection and orally on Day 16.
- Group 2: Moxifloxacin 400mg: Participants received a single oral dose of 400 mg moxifloxacin on Day 10.
- Group 3: Placebo: Participants received once daily Placebo from Days 1 to 16, via SC injection and orally on Day 10.
- Group 3: Moxifloxacin 400mg: Participants received a single oral dose of 400 mg moxifloxacin on Day 16.
Arm/Group | Group 1: Setmelanotide 2 mg | Group 1: Setmelanotide 3 mg | Group 1: Setmelanotide 5 mg | Group 1: Setmelanotide 7 mg | Group 2: Placebo | Group 2: Moxifloxacin 400mg | Group 3: Placebo | Group 3: Moxifloxacin 400mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/24 | 0/23 | 0/21 | 0/24 | 0/23 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/24 | 0/23 | 0/21 | 0/24 | 0/23 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 25/28 | 16/24 | 17/23 | 9/21 | 18/24 | 17/23 | 15/25 | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Setmelanotide 2 mg (N=28) | Group 1: Setmelanotide 3 mg (N=24) | Group 1: Setmelanotide 5 mg (N=23) | Group 1: Setmelanotide 7 mg (N=21) | Group 2: Placebo (N=24) | Group 2: Moxifloxacin 400mg (N=23) | Group 3: Placebo (N=25) | Group 3: Moxifloxacin 400mg (N=25)
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Setmelanotide 2 mg (N=28) | Group 1: Setmelanotide 3 mg (N=24) | Group 1: Setmelanotide 5 mg (N=23) | Group 1: Setmelanotide 7 mg (N=21) | Group 2: Placebo (N=24) | Group 2: Moxifloxacin 400mg (N=23) | Group 3: Placebo (N=25) | Group 3: Moxifloxacin 400mg (N=25)
Injection site pain (General disorders) | 11 | 7 | 6 | 7 | 8 | 12 | 11 | 0
Injection site erythema (General disorders) | 7 | 10 | 7 | 2 | 1 | 6 | 6 | 0
Injection site pruritus (General disorders) | 3 | 4 | 3 | 1 | 3 | 1 | 4 | 0
Injection site swelling (General disorders) | 4 | 1 | 3 | 4 | 1 | 4 | 9 | 0
Fatigue (General disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Medical device site dermatitis (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1
Injection site bruising (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0
Injection site discolouration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 0 | 4 | 2 | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 8 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival discolouration (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lip discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pigmentation lip (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue pigmentation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 6 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Allodynia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erection increased (Reproductive system and breast disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in sexual arousal (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT05046132/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT05046132/SAP_002.pdf